CLINICAL TRIAL: NCT02113163
Title: An Open-label, Single and Repeat Single Ascending Dose Escalation Study to Compare the Pharmacokinetics of Metformin Eicosapentaenoate With Metformin Hydrochloride and Icosapent Ethyl Following Oral Administration to Healthy Volunteers
Brief Title: PK Study Comparing Metformin Eicosapentaenoate to a Combined Dose of Metformin Hydrochloride and Ethyl Ester EPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thetis Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-101-CS01
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Hypertriglyceridemia
Keywords: Type 2 diabetes; T2DM; hypertriglyceridemia; severe hypertriglyceridemia; dyslipidemia; triglycerides; lipids; omega-3 fatty acids; EPA; ethyl-EPA; Metformin; Glucophage; Lovaza; Vascepa; Epanova; Astra Zeneca; Amarin; GSK
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertriglyceridemia; Dyslipidemias | interventions — Metformin; eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A - Low Dose (Active Comparator): Metformin Eicosapentaenoate 1500 mg or Metformin HCl 500 mg and Vascepa 1000 mg
  Interventions: Drug: Metformin Eicosapentaenoate; Drug: Metformin HCl and Vascepa
- Cohort B - High Dose (Active Comparator): Metformin Eicosapentaenoate 3000 mg or Metformin HCl 1000 mg and Vascepa 2000 mg
  Interventions: Drug: Metformin Eicosapentaenoate; Drug: Metformin HCl and Vascepa

INTERVENTIONS:
Drug: Metformin Eicosapentaenoate
Drug: Metformin HCl and Vascepa

SUMMARY:
The primary objective of the study is to contrast the pharmacokinetic profiles of metformin and EPA delivered separately as co-administered products (metformin hydrochloride or Glucophage and icosapent ethyl or Vascepa) and together as the solid dose form (metformin eicosapentaenoate or TP-101) under fasted and fed conditions. A secondary objective is to evaluate the safety and tolerability of single and repeat single doses of TP-101.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent executed prior to protocol screening assessments;
* Men or women 18 to 65 years of age, inclusive (Women may be surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are postmenopausal for >1 year. Women who are of childbearing potential must agree to practice adequate contraception one month before the first dose of study medication and up to Day 16 of the study. Adequate contraception may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms or diaphragms with spermicide or foam, intrauterine devices, and licensed hormonal methods.);
* No history of chronic diseases, except for subjects with well-controlled hypertension or well-controlled hyperlipidemia;
* BMI ≤30kg/m2;
* No significant medical history including diabetes or hypertension complicated by hyperlipidemia (metabolic syndrome);
* Negative urine drug and alcohol tests at Screening; and,
* No metformin or omega-3 products within 2 months.

Exclusion Criteria:

* Abnormal findings on physical examination, EKG, vital signs, and clinical laboratory testing, in the judgment of the investigator;
* Allergies to fish or shellfish;
* Impaired renal function (calculated eGFR <60 mL/min);
* Abnormal laboratory values for T3, T4 and TSH at the Screening Visit;
* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) >2x upper limits of normal (ULN) or serum bilirubin >1.5 mg/dL;
* Requirement of prescription medication within 14 days of the Screening Visit, with the exception of prescription medications for the prevention of pregnancy, anti hypertensives for hypertension, or statins for hyperlipidemia. Doses of one or two anti-hypertensives and/or a statin must be stable for >1 month;
* Normal doses of over-the-counter medications, including vitamins are allowed but not within 3 days of Visit 2 (first day of dosing);
* Current or history of abuse of alcohol or illicit drugs within the preceding year to the Screening Visit;
* Participation in a dietary modification or an intensive weight loss program;
* Participation in another clinical trial of an investigational product within 3 months prior to the Screening Visit;
* Smokers (use of tobacco in the past 3 months); or,
* Donation or loss of 400 mL blood or more in the last 8 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
AUC following single and repeat single oral administration of metformin eicosapentaenoate, metformin hydrochloride and Vascepa | PK samples at 0, 0.5, 1, 2, 4, 8, and 12 hours following drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States